CLINICAL TRIAL: NCT06865872
Title: Alcohol and Sexual Communication Among Couples in the Laboratory
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-1867; R01AA031666 (NIH)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Intoxication; Intimate Partner Violence (IPV); Communication
MeSH Terms: conditions — Alcoholic Intoxication; Communication | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcohol Consumption + Direct Communication (Experimental): Participants will be assigned to drink alcohol and to receive direct communication about their sexual preferences from their partner.
  Interventions: Other: Direct Communication; Drug: Alcohol (Ethanol)
- Alcohol Consumption + Indirect Communication (Experimental): Participants will be assigned to drink alcohol and to receive indirect communication about their sexual preferences from their partner.
  Interventions: Other: Indirect Communication; Drug: Alcohol (Ethanol)
- No Alcohol + Direct Communication (Experimental): Participants will be assigned to drink a no-alcohol control beverage and to receive direct communication about their sexual preferences from their partner.
  Interventions: Other: Direct Communication; Other: No-Alcohol Control
- No Alcohol + Indirect Communication (Experimental): Participants will be assigned to drink a no-alcohol control beverage and to receive indirect communication about their sexual preferences from their partner.
  Interventions: Other: Indirect Communication; Other: No-Alcohol Control

INTERVENTIONS:
Other: Direct Communication — Participants assigned to receive direct communication about their sexual preferences from their partner.
  Arms: Alcohol Consumption + Direct Communication; No Alcohol + Direct Communication
Other: Indirect Communication — Participants assigned to receive indirect communication about their sexual preferences from their partner.
  Arms: Alcohol Consumption + Indirect Communication; No Alcohol + Indirect Communication
Drug: Alcohol (Ethanol) — Participants assigned to moderate alcohol dose condition (target BrAC .10%) with the National Institute on Alcohol Abuse and Alcoholism (NIAAA) approved alcohol administration procedures.
  Arms: Alcohol Consumption + Direct Communication; Alcohol Consumption + Indirect Communication
Other: No-Alcohol Control — Participants assigned to a no-alcohol control beverage.
  Arms: No Alcohol + Direct Communication; No Alcohol + Indirect Communication

SUMMARY:
Intimate Partner Sexual Violence (IPSV) is a significant and understudied public health problem among couples, yet little is known about factors that contribute to IPSV perpetration. This proposal aims to determine the acute effect of alcohol and sexual communication on IPSV. In this study, 240 couples who drink alcohol will be recruited from the Metro-Denver area. Upon arrival to the laboratory, a trained research assistant will check the participant's ID, verify that they adhered to the pre-session guidelines, administer a breath test to ensure a breath alcohol content (BrAC) of 0.00 and conduct a field sobriety test. They will also obtain informed consent for each member of the couple separately. Female participants will take a pregnancy test to ensure a negative result. All participants will complete measures to reverify eligibility criteria and be weighed to determine their correct alcohol dose. Partners will separately complete a baseline survey measuring demographic factors, alcohol use, sexual communication, and daily experiences. After completing the survey, participants will be assigned a beverage condition (alcohol or no-alcohol control) and couples will be randomly assigned to a communication condition (direct verbal or indirect verbal). Participants will be seated in a room separate from their partner, where they will drink an alcoholic or no-alcohol control beverage. Upon reaching a breath alcohol content (BrAC) of .07, or immediately after drinking in the No-Alcohol control condition, participants will complete a laboratory assessment of sexual violence. The main hypotheses are: (1) one's alcohol use will increase IPSV toward partners who are also drinking, (2) one's alcohol use will increase IPSV among partners who use indirect, relative to direct, communication, and (3) actor alcohol use will increase IPSV toward partners who are also drinking and use indirect, relative to direct, communication.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and lifestyle considerations.
3. Both partners must identify as cisgender via self-report on the Baseline Questionnaire.
4. At least one partner within the couple must be a man via self-report on the Baseline Questionnaire.
5. Both partners must be between 21 and 65 years old, verified by a photo ID.
6. In an intimate relationship lasting at least one month in which they engaged in sexual activity at least once in the past month with their partner via self-report on the Baseline Questionnaire.
7. Both partners must report that they consumed a weight-based amount of alcohol that is equal to or greater than the dose to be administered in the lab at least three times during the past year via self-report on question #5 of the NIAAA Alcohol Consumption Measure.

Please contact clinical site for additional inclusion criteria.

Exclusion Criteria:

1. Treatment for Alcohol or Drug Use: currently being treated for alcohol, or drug problems; currently interested in seeking treatment for drinking or drug use via self-report.
2. Any medical or psychiatric condition, as well as current use of a medication, that would contraindicate alcohol administration via self-report:

   * Cardiac Pacemaker
   * Asthma: emergency room visit related to asthma in the past year; use of inhaler more frequently when drinking alcohol; use of oral steroid treatments for asthma in the past year
   * Head Injury: any past serious head injuries
   * Acute Psychiatric Symptomatology: elevated psychological distress as indicated by a score greater than 65 on the Brief Symptom Inventory
3. Self-report that a participant is trying to get pregnant, currently pregnant, or currently breastfeeding or a positive pregnancy test.
4. Combined height and weight that is either less than 6 feet tall and over 230 lbs, or over 250 lbs and over 6 ft tall as measured during the lab visit.

Please contact clinical site for additional exclusion criteria.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both partners must identify as cisgender and at least one partner must identify as a man.
Enrollment: 480 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Sexual Violence Perpetration as Measured by the Sexual Imposition Paradigm | up to 1 hour post beverage consumption
  The Sexual Imposition Paradigm measures sexual violence perpetration. Possible scores are 0 (no perpetration) to 1 (perpetration).
Sexual Violence Perpetration Length of Time as Measured by the Sexual Imposition Paradigm | up to 1 hour post beverage consumption
  The Sexual Imposition Paradigm measures sexual violence perpetration length of time. Scores range from 0 to 120 seconds, with higher scores indicating longer perpetration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available in the NIAAA Data Archive.